CLINICAL TRIAL: NCT05321589
Title: Accuracy of Digital and Conventional Impression Techniques for Maxillary Full Arch Screw Retained Hybrid Prosthesis
Brief Title: Accuracy of Conventional and Digital Impression Techniques Used for Maxillary Hybrid Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Gilan Altonbary, associate professor, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A25100221
Record Dates: First submitted 2022-03-21; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Prosthesis Durability
Keywords: digital impression, conventional impression
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: the conventional open tray splinted impression technique and the digital intraoral impression technique were done for each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- technique 1: conventional splinted open tray impression (Other): a conventional open tray impression technique splinted with ligature wire and duralay resin was done with polyvinyl siloxane impression .
  analogues were screwed to the impression copings and casts were poured.
  Interventions: Other: impression techniques for implant used for maxillary screw retained hybrid prosthesis
- technique 2: digital intraoral impression technique (Other): scan bodies were screwed to implants intraorally and digital scanner was used to record digital impression, scanning protocol started from occlusal ,buccal to palatal surfaces.
  The resulting scans were then exported in the standard tessellation format (.STL)
  Interventions: Other: impression techniques for implant used for maxillary screw retained hybrid prosthesis

INTERVENTIONS:
Other: impression techniques for implant used for maxillary screw retained hybrid prosthesis — conventional splinted open tray impression technique was done for maxillary implants to fabricate screw retained hybrid prosthesis and digital intra oral impression was done for the same patients after screwing scan bodies to the implants intra orally.
  evaluation of accuracy and 3D deviation between the two techniques was done
  Other Names: digital and conventional impression techniques

SUMMARY:
evaluation and comparison of the accuracy of conventional and digital impression for full arch screw retained prosthesis for edentulous maxilla.

DETAILED DESCRIPTION:
Each patient received 6 implants in the maxillary ridge (widely distributed across the arch) in the following positions: central incisors, canines/first premolar teeth and first molar teeth aided by surgical stent. then each patient received 2 types of impression techniques Technique 1 :conventional impression conventional open tray impression technique with splinted transfers using vinylpolysiloxane and Technique2 : Digital impression taken using original scan bodies torqued to the implants .three dimensional accuracy of impression techniques was evaluated using linear measurements and 3D deviation between the two techniques was measured.

ELIGIBILITY:
Inclusion Criteria:

* The patients were selected according to the following inclusion criteria:

  1. Completely edentulous maxillary and mandibular ridges
  2. Healthy ridge covered by normal oral mucosa and free from any ridge flabbiness.
  3. All of the patients were dissatisfied with the retention and stability of their maxillary conventional dentures and expressed a strong desire for a more stable prosthesis.
  4. Sufficient bone quantity and quality in the front and posterior maxillary regions, as determined by preoperative CBCT, to accommodate six implants with a diameter of at least 3.5 mm and a length of at least 10 mm.
  5. Enough restorative space (from the mucosa covering the crest of the maxillary residual ridge to the occlusal plane) to allow the fixed prosthesis to be constructed ,preliminary jaw relationship revealed this.
  6. It's been at least a year since the last extraction.

     Exclusion Criteria:

  <!-- -->

  1. Systemic diseases that may alter tissue response to implantation and affects osseointegration (radiation, diabetes, osteoporosis, bleeding disorders or hepatic patients)
  2. Long term immunosuppressive and corticosteroid drug therapy.
  3. Patient with abnormal habits as clenching and bruxism.
  4. Smoking patients.
  5. Patients with problems in TMJ.
  6. Neuromuscular diseases.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
accuracy of impression technique | immediately after the intervention/procedure
  deviation measurements digitally

SECONDARY OUTCOMES:
passivity of final restoration | immediately after the intervention/procedure
  Clinical measurement of prosthesis passivity using single screw test of Sheffield.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of Dentistry , Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No